CLINICAL TRIAL: NCT06072521
Title: Efficacy of Lactoferrin as an Adjunct Therapy in Patients With Hepatic Encephalopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Kholoud El-Sayed Ibrahim, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Lactoferrin in HE
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled clinical trial (Pilot study) that will be conducted on hepatic encephalopathy patients who will attend to National Hepatology and Tropical Medicine Research Institute, Cairo, Egypt to receive the treatment regimen in concurrence with the Egyptian guidelines of treatment. Eligible patients will randomly assigned in a 1:1:1 ratio to receive lactoferrin (Pravotin@ sachets) as followings:
  Group I: Patients receive standard care alone (control group) Group II: Patients receive 100mg lactoferrin orally (one sachet (100 mg), one time a day) plus standard care.
  Group III: Patients receive 200 mg lactoferrin orally (one sachet (100mg), two times a day) plus standard care. Lactoferrin will be administrated in groups II and III for 15 days. The blood samples of all eligible participants and reported signs and symptoms will be collected after 15 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lactoferrin bovine once a day (Active Comparator): 15 patients will be subjected to take 100mg of lactoferrin bovine in the form of sachets twice per day for 15 days.
  Interventions: Drug: Lactoferrin Bovine
- Lactoferrin bovine twice a day (Active Comparator): 15 patients will be subjected to take 100mg of lactoferrin bovine in the form of sachets once per day for 15 days.
  Interventions: Drug: Lactoferrin Bovine
- Control group (No Intervention): 15 patients will be subjected to take only the standard treatment regimen that is applied at the National hepatology and tropical medicine research institute in Egypt.

INTERVENTIONS:
Drug: Lactoferrin Bovine — Lactoferrin bovine with concentration 100 mg will be given to the patients in test groups in the form of sachets.
  Other Names: Pravotin sachets 100 mg
  Arms: Lactoferrin bovine once a day; Lactoferrin bovine twice a day

SUMMARY:
The aim of this study is to evaluate the efficacy of lactoferrin as an adjunct therapy in improving clinical symptoms and laboratory indices in individuals with hepatic encephalopathy.

DETAILED DESCRIPTION:
Nonabsorbable disaccharides, such as lactulose or lactitol, decrease the absorption of ammonia and are considered a first-line treatment for hepatic encephalopathy. Antimicrobial therapy also is a part of treatment regimen to alter the gut microbiota to create a more favorable microbiome that results in lower endogenous bacterial production of ammonia and Rifaximin is now the preferred antimicrobial agent for the treatment of hepatic encephalopathy. Many researchers have focused on identifying promising therapeutics and prebiotics in the hope of improving the treatment of hepatic encephalopathy, therefore there is a need to add an adjuvant therapy to decrease oxidative stress and pro-inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Grade I and II hepatic encephalopathy.

Exclusion Criteria:

* Pregnant and breastfeeding women.
* Grade III and IV hepatic encephalopathy.
* Individuals confirmed to be allergic to milk protein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in serum concentration of inflammatory cytokines | 15 days
  Change in serum concentration of inflammatory cytokine Tumor necrosis factor-alpha (TNF-a) (pg/ml)
Change in serum concentration of Nuclear factor kB | 15 days
  Change in serum concentration of Nuclear factor kB (NFkB) (ng/ml)
Change in serum concentration of oxidative stress markers | 15 days
  Change in serum concentration of oxidative stress markers Malondialdehyde (MDA) (n.mol/mg/protein) and Glutathione (GSH) (m.mol/mg/protein)

SECONDARY OUTCOMES:
Change in Psychometric Hepatic Encephalopathy Score (PHES) | 15 days
  Number connection test A (NCT-A) - in this test the numbers have to be joined consecutively in ascending numerical order (1, 2, 3…) as quickly as possible.
Change in Psychometric Hepatic Encephalopathy Score (PHES) | 15 days
  Digit symbol test (DST) - in this test the patient is given a series of double-boxes with a number given in the upper part. The task is to draw a symbol pertinent to this number into the lower part of the boxes. Nine fixed pairs of numbers and symbols are given at the top of the test sheet. Test result is the number of boxes correctly filled within 90 seconds.
Change in Psychometric Hepatic Encephalopathy Score (PHES) | 15 days
  Simplified animal naming test (S-ANT) - in this test patients are asked to name as many animals as possible in one minute. Repeats and errors were excluded from the calculation. The number of named animals after one minute was the definitive score.
Length of hospital stay | 15 days
  Length of hospital stay
The rate of adverse events occurring during the treatment | 15 days
  Number of patients who experienced adverse events such as diarrhea, rash, loss of appetite, fatigue, and constipation.
Number of patients transferred to ICU | 15 days
  Number of patients transferred to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Amin M. Abdel Baki, Doctoral, Study Chair — National hepatology and tropical medicine research institute; Nayira A. Abdel Baky, Doctoral, Study Director — Al-Azhar University
Locations (1):
- National hepatology and tropical medicine research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bajaj JS. Hepatic encephalopathy: classification and treatment. J Hepatol. 2018 Apr;68(4):838-839. doi: 10.1016/j.jhep.2017.11.005. No abstract available. PMID 29756596
- [Background] Patidar KR, Bajaj JS. Covert and Overt Hepatic Encephalopathy: Diagnosis and Management. Clin Gastroenterol Hepatol. 2015 Nov;13(12):2048-61. doi: 10.1016/j.cgh.2015.06.039. Epub 2015 Jul 9. PMID 26164219
- [Background] Elsaid MI, Rustgi VK. Epidemiology of Hepatic Encephalopathy. Clin Liver Dis. 2020 May;24(2):157-174. doi: 10.1016/j.cld.2020.01.001. Epub 2020 Mar 2. PMID 32245524